CLINICAL TRIAL: NCT00383526
Title: Study of Inactivated, Split-Virion Influenza Vaccine Compared With the Reference Vaccine Vaxigrip® in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GID17
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine; elderly
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group 1 (Experimental)
  Interventions: Biological: Inactivated, split-virion influenza vaccine
- Study Group 2 (Active Comparator)
  Interventions: Biological: Inactivated, split-virion influenza vaccine

INTERVENTIONS:
Biological: Inactivated, split-virion influenza vaccine — Vaccine
  Arms: Study Group 1
Biological: Inactivated, split-virion influenza vaccine — Vaccine
  Other Names: Vaxigrip®
  Arms: Study Group 2

SUMMARY:
Vaccination against influenza is a high priority for the elderly population who present the highest morbidity and mortality rate. However, due to their weak antibody response an improvement of the immune response to influenza vaccination remains an unmet medical need. The purpose of an investigational influenza vaccine candidate administered by an alternate route is to improve immune responses to the vaccine in the elderly population, which could provide additional reductions in influenza-associated morbidity and mortality in this population.

Primary Objective:

To demonstrate that the investigational vaccine induces a better immunogenicity than the reference vaccine in terms of seroprotection rate after the first vaccination.

Secondary Objectives:

Immunogenicity:

To describe the antibody persistence induced by both vaccines at 3, 6, and 12 months after the first vaccination in a subset of subjects.

To describe the immunogenicity of the investigational vaccine after each vaccination using parameters defined in the European Medicines Agency (EMEA) Note for Guidance (CPMP/BWP/214/96) specific to elderly subjects.

Safety:

To demonstrate the tolerance of the investigational vaccine after the first vaccination, in terms of pre-defined solicited systemic reactions.

To describe the safety profile after each vaccination. To describe the effect of repetitive injections on the safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 60 years on the day of inclusion.
* Informed Consent Form signed.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Systemic hypersensitivity to egg proteins, chick proteins, or any of the vaccine components, in particular, neomycin, formaldehyde, and octoxinol 9, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Febrile illness (oral temperature ≥ 37.5°C or rectal equivalent temperature ≥ 38.0°C) on the day of inclusion.
* Participation in another clinical trial in the four weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Unstable chronic illness (defined as illness requiring hospitalization or a clinically significant change in medication in the 12 weeks prior to inclusion) at a stage that could interfere with trial conduct or completion.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Blood or blood-derived products received in the past 3 months.
* Any vaccination in the 4 weeks preceding the first trial vaccination.
* Vaccination planned in the 4 weeks following the first trial vaccination.
* Previous vaccination against influenza (in the previous 6 months) with the trial vaccine or another vaccine.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3707 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of Inactivated, Split-Virion Influenza vaccine | 21 days post-vaccination

SECONDARY OUTCOMES:
To provide information concerning the safety of Inactivated, Split-Virion Influenza vaccine | Entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (4):
- Antwerp, Belgium
- Angers, France
- Genova, Italy
- Vilnius, Lithuania

REFERENCES:
- [Derived] Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection (VAPI) questionnaire. Health Qual Life Outcomes. 2009 Mar 4;7:21. doi: 10.1186/1477-7525-7-21. PMID 19261173
- See also: Related Info — http://www.sanofipasteur.com